CLINICAL TRIAL: NCT04423744
Title: Randomized, Single-blind, Double-dummy, 4-fold Cross-over, Placebo- and Active-controlled Study to Investigate the Influence of BAY 1817080 on the QTc Interval in Healthy Male and Female Participants (TQT Study)
Brief Title: Study to Gather Information on the Influence of BAY1817080 on the Electrical Activity of the Heart Recorded by an Electrocardiogram in Healthy Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 21198; 2020-000516-29 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Cough; Endometriosis; Overactive Bladder
MeSH Terms: conditions — Cough; Endometriosis; Urinary Bladder, Overactive | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention ABCD (Experimental): Intervention A:
  Day 1 and 2: Supra-therapeutic dose of BAY1817080, three times daily (tid) Day 3: Supra-therapeutic dose of BAY1817080 and placebo to moxifloxacin, once
  Intervention B:
  Day 1 and 2: therapeutic dose of BAY1817080 and placebo to BAY1817080, tid Day 3: therapeutic dose of BAY1817080, placebo to BAY1817080 and placebo to moxifloxacin, once
  Intervention C:
  Day 1 and 2: Placebo to BAY1817080, tid Day 3: Placebo to BAY1817080 and moxifloxacin, once
  Intervention D:
  Day 1 and 2: Placebo to BAY1817080, tid Day 3: Placebo to BAY1817080 and placebo to moxifloxacin, once
  Subjects will receive intervention A, B, C and D sequentially. The washing-out period between each intervention is at least 14 days
  Interventions: Drug: BAY1817080; Drug: Moxifloxacin; Drug: Placebo
- Intervention BCDA (Experimental): Subjects will receive intervention B, C, D and A sequentially. The washing-out period between each intervention is at least 14 days
  Interventions: Drug: BAY1817080; Drug: Moxifloxacin; Drug: Placebo
- Intervention CDAB (Experimental): Subjects will receive intervention C, D, A and B sequentially. The washing-out period between each intervention is at least 14 days
  Interventions: Drug: BAY1817080; Drug: Moxifloxacin; Drug: Placebo
- Intervention DABC (Experimental): Subjects will receive intervention D, A, B and C sequentially. The washing-out period between each intervention is at least 14 days
  Note: the intervention sequences in this and above arms are examples, the actual order of intervention may differ from these examples
  Interventions: Drug: BAY1817080; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: BAY1817080 — Film-coated tablet
Drug: Moxifloxacin — Film-coated tablet
Drug: Placebo — Matched placebo as film-coated tablet

SUMMARY:
In this study, researchers want to find whether the study drug BAY1817080 has an effect on the electrocardiogram (ECG). 40 healthy male or female participants with the age of 18 to 65 years will be enrolled into this study. The ECG of the participants will be monitored closely by the researchers to detect any change after intake of the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Men must be 18 to 65 years of age inclusive, women must be 40 to 65 years of age inclusive at the time of signing the informed consent
* Female participants have to be in postmenopausal state
* Body mass index (BMI) within the range 18.0-32.0 kg/m^2 (inclusive)
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, ECG, and vital signs
* 12-lead electrocardiogram recording without signs of clinically relevant pathology

Exclusion Criteria:

* A history of relevant diseases of vital organs, of the central nervous system or other organs
* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention will not be normal
* Known hypersensitivity to the study interventions (active substances, or excipients of the preparations)
* Known severe allergies e.g. allergies to more than 3 allergens, allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids, urticaria or significant nonallergic drug reactions
* Febrile illness within 1 week before study intervention administration
* Known or suspected disorder of the liver (e.g. bile secretion/flow disorder, Morbus Meulengracht (Gilbert´s syndrome), drug-induced hepatitis etc.)
* History of disorder of the pancreas or evidence for past or present pancreas disorders indicated by clinically relevant lipase or amylase levels above ULN and typical clinical symptoms of pancreas disorders as e.g. upper abdominal pain spread to the back, weight loss, fatty or pale stools
* Participants with thyroid disorders as evidenced by assessment of thyroid stimulating hormone (TSH) levels outside the normal reference range at screening (inclusion with normal fT3/fT4 levels allowed)
* History of known or suspected malignant tumors
* History of hypokalemia
* Use of CYP3A4 inhibitors from 14 days before study intervention administration until the last study visit
* Use of CYP3A4 inducers within 4 weeks (or at least five half-lives of the active substance whatever is longer) prior to study intervention administration
* Smoking more than 10 cigarettes daily
* Suspicion of drug or alcohol abuse
* Plasmapheresis within 3 months prior to study drug administration
* Excluded physical therapies that might alter the PK or safety results of the study (e.g. physiotherapy, acupuncture, etc.) from 7 days before first study drug administration until follow-up
* Systolic blood pressure below 100 mmHg or above 140 mmHg at screening. Difference of systolic BP between both arms >15 mmHg
* Diastolic blood pressure below 50 mmHg or above 90 mmHg at screening
* Heart rate below 50 beats/ min or above 90 beats/ min at screening
* History of COVID-19
* Prior contact with SARS-CoV-2 positive or COVID-19 patient within the last 4 weeks prior admission to the ward
* Positive SARS-CoV-2 viral test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Time-matched, placebo-corrected change from baseline of the individually corrected QT interval after multiple oral doses of BAY1817080 therapeutic dose | Baseline and Day 3
Time-matched, placebo-corrected change from baseline of the individually corrected QT interval after multiple oral doses of BAY1817080 supra-therapeutic dose | Baseline and Day 3

SECONDARY OUTCOMES:
Time-matched, placebo-corrected change from baseline of the individually corrected QT interval after a single oral dose of moxifloxacin | Baseline and Day 3
Time-matched, placebo-corrected change from baseline of the QT interval corrected according to Fridericia (QTcF) and Bazett (QTcB) after multiple oral doses of BAY1817080 therapeutic or supra-therapeutic dose | Baseline and Day 3
Time-matched, placebo-corrected change from baseline of the QT interval corrected according to Fridericia (QTcF) and Bazett (QTcB) after a single oral dose of moxifloxacin | Baseline and Day 3
AUC(0-24)md after multiple oral doses of BAY1817080 therapeutic or supra-therapeutic dose | Predose and up to 24 hours after last dose of BAY1817080 at Day 3
  Area under the concentration vs. time curve from zero to 24 hours after multiple doses
AUC after a single oral dose of moxifloxacin | Predose and up to 24 hours after single dose of moxifloxacin at Day 3
  Area under the concentration vs. time curve from zero to infinity after single dose
Cmax,md after multiple oral doses of BAY1817080 therapeutic or supra-therapeutic dose | Up to 24 hours after last dose of BAY1817080 at Day 3
  Maximum observed drug concentration in measured matrix after multiple doses
Cmax after a single oral dose of moxifloxacin | Up to 24 hours after single dose of moxifloxacin at Day 3
  Maximum observed drug concentration in measured matrix after single dose
Incidences of treatment-emergent adverse events (TEAEs) after BAY1817080 therapeutic or supra-therapeutic dose | From the start of BAY1817080 administration until 7 days after last dose, assessed up to 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.